CLINICAL TRIAL: NCT05766436
Title: Nebulized Dexmedetomidine VS Oro-dispersible Film Melatonin for Peri Operative Anxiety and Emergence Agitation in Pediatric Outpatient Surgeries: A Randomized Controlled Double-blinded Study
Brief Title: Nebulized Dexmedetomidine VS ODF Melatonin for Peri Operative Anxiety and Emergence Agitation in Pediatric Day Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: nada moahmed aboelrouse (Other)
Responsible Party: Sponsor-Investigator, nada moahmed aboelrouse, assistant lecturer, NewGiza University
Organization: NewGiza University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWA 000017585
Record Dates: First submitted 2023-02-19; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Anxiety Acute; Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Melatonin; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group D (Active Comparator): will receive placebo ODF and nebulized dexmedetomidine (Precedex™ rxlist)
  Interventions: Drug: Dexmedetomidine
- group M (Active Comparator): will receive placebo nebulizer and ODF melatonin (metacyst ™ nerhadou)
  Interventions: Drug: Melatonin
- group C (Placebo Comparator): will receive placebo ODF and placebo 0.9% normal saline nebulizer
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — receive placebo ODF and 3 µ/kg nebulized dexmedetomidine (Precedex™ rxlist) prepared in 0.9% normal saline to a final volume of 3ml. Nebulization was performed using a wall nebulizer and wall oxygen source on 4 l/min.
  Other Names: Precedex™ rxlist
  Arms: group D
Drug: Melatonin — will receive placebo nebulizer and 0.4mg/kg of ODF melatonin (metacyst ™ nerhadou) orally allowing the film to dissolve in the patients Oro mucosal lining
  Other Names: metacyst ™ nerhadou
  Arms: group M
Drug: Placebo — placebo ODF and 0.9% normal saline nebulizer
  Other Names: normal saline
  Arms: group C

SUMMARY:
The goal of this clinical trial is to compare between the effect of nebulized dexmedetomidine and the effect of oral dispensable film (ODF) melatonin in controlling perioperative anxiety and post operative emergence agitation and their effect on the overall surgical experience.in pediatric patients undergoing day case surgery.

DETAILED DESCRIPTION:
All patients will be admitted on the day of the surgery and will be instructed to fast 6 hours before surgery for older patients, as for breast fed patients, they will be instructed for 4 hours for breast feeding and for formula fed patients they will be instructed to fast for 6 hours as recommended by the American society of anesthesiologists. Preoperative assessment will be done before surgery by one of the members of the team who will make sure that the inclusion and exclusion criteria of the patients are considered, and baseline vital signs will be recorded. According to randomization that will be done by envelop concealed allocation , the drug will be administered to the patients by a researcher who will not participate in the evaluation of the patients 30 mins before transfer to the operation room (OR): each group will receive the intervention drug Parents are not allowed to accompany their children to the OR according to the hospital policy. On arrival to the OR department the Parental separation anxiety scale (PSAS) will be calculated on entering the operation room standard monitoring will be commenced including ECG, non-invasive blood pressure and pulse oximetry and baseline measurement will be recorded. Inhalational induction will be then started with sevoflurane and mask acceptance will be calculated according to the mask acceptance scale (MAS) intravenous cannulation will be then established after which each patient will receive 1-2 mg/kg Propofol, 1 µg/kg fentanyl to attenuate the stress of intubation and 0.5mg/kg atracurium after tracheal intubation anesthesia will be maintained with sevoflurane 2-4 MAC During the length of the operation vital data will be recorded at 5 minutes interval. all patients will receive IV paracetamol 15mg/kg and patient would receive 1 µg/kg fentanyl as a rescue dose if vital data increased by >20% of the baseline.

after the completion of surgery extubating will be performed after meeting extubation criteria and patient will be discharged to post-anesthesia care unit (PACU) in for the first 15 min after admission to PACU the post anesthesia emergence agitation will be assessed by using Pediatric Anesthesia Emergence Delirium Scale (PAED) during the stay in PACU pain will also be assessed by using FLACC score Discharge from PACU will be done after meeting discharge criteria and the time of discharge will be documented. After discharge pain score will be measured using FLACC score at 15, 30, 60 minutes interval postoperative and the total combustion of postoperative analgesics will be calculated as well as the time of discharge from the hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists (ASA) physical status I & II
* both genders,
* ≥ 2 to 10 years,
* scheduled for elective day case surgery under general anesthesia

Exclusion Criteria:

* parents' refusal for participation in the study
* ASA III and VI patients with history of chronic illness
* runny nose or upper respiratory tract infection
* Emergency surgeries with hemodynamic instability
* history of allergic reaction to dexmedetomidine or melatonin
* History of prematurity
* developmental delay
* central nervous system disorder,
* mental retardation,
* neurological or psychiatric illness that may be associated with anxiety and agitation (cerebral palsy, seizure, separation anxiety disorder, ADHD etc.).
* treatment with anticonvulsants and sedatives

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
perioperative anxiety | during the patient separation from the caregiver just as the child is going to the operating theater
  perioperative anxiety will be measured by using Parental separation anxiety scale (PSAS) will be calculated according to the following:
  * Behavior of the child during separation from parents will be Excellent if the Patient unafraid, cooperative, or asleep will be given the score of (1)
  * Behavior of the child during separation from parents will be Good if the patient is Slightly afraid/crying, quiet with reassurance will be given the score (2)
  * Behavior of the child during separation from parents will be Fair if the patient is Moderately afraid and crying not quit with reassurance with the score (3)
  * Behavior of the child during separation from parents will be poor if the patient is Crying, need for restraint with the score (4)
  the score of (1) means excellent response , score of (2) means good response , score of (3) means fair response and score of (4) means poor response

SECONDARY OUTCOMES:
mask acceptance | during the mask introduction to start inhalational induction of anesthesia with sevoflurane before skin incision
  calculated according to the mask acceptance scale (MAS) as following : if the Child is calm, cooperative, or asleep the score will be (1) if the child is in Moderate fear of the mask Manageable with reassurance the score will be(2) if the child Cries, combative and needs restraining the score will be (3)
  score of (1) means excellent response ,score of (2) means fair response and score of (3) means poor response
post anesthesia emergence agitation | first 15 minutes after admission to post- anesthesia care unit
  will be assessed by using Pediatric Anesthesia Emergence Delirium Scale (PAED) with score
  1= calm , 2= not calm but could be easily consoled , 3= moderately agitated or restless and not easily calmed , 4 = combative , excited , thrashing around
pain score | during hospital stay up to 3 hours
  using Face, leg, activity, cry and Consolability score With score of 0 meaning no pain and requires no intervention and score of 10 indicating the worst imaginable pain requiring rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Sohair Abbas, MD, Study Chair — Ain Shams University, Anesthesia department; Ramy Mahrose, MD, Study Director — Ain Shams University, Anesthesia department; Wessam Zaher, MD, Study Director — Ain Shams University, Anesthesia department
Locations (1):
- Ain shams university hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No